CLINICAL TRIAL: NCT02310217
Title: Validation of New Tools for the Assessment of Cognitive Functions and Connectivity Network in Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB03
Record Dates: First submitted 2014-11-28; First posted 2014-12-08 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Hypertension; Cognitive Impairment
Keywords: Hypertension; Cognitive impairment; Biomarkers
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 1: Hypertensive
- 2: Normotensive

SUMMARY:
The relationship among hypertension, aging and cognitive decline is complex and not completely understood. Purpose of this project will be evaluating early markers of cognitive deterioration in patients with arterial hypertension. In particular, this cross-sectional observational study will be articulated in three phases:

1. Neuropsychological evaluation of general cognitive abilities
2. Identification and measurement of specific biomarker levels
3. Correlation among hypertension, cognitive abilities and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Males or females diagnosed with arterial hypertension between 40 and 65 years of age;
* Written informed consent prior to enrollment in the study.

Exclusion Criteria:

* Precedent acute myocardial infarction (AMI);
* Previous stroke and/or transient ischemic attack (TIA);
* Previous or concomitant neurologic or psychiatric pathologies;
* Neurologic or psychiatric pharmacological therapy.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Department of Angiocardioneurology and Translational Medicine of the IRCCS Neuromed, according to specific inclusion criteria. Approximatey 80 subjects per group, aged between 40 and 65 years, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Cognitive abilities measured by validated neuropsychological test battery (Montreal Cognitive Assessment test, Verbal Fluency test,learning of couple words, Stroop test) | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, (IS), Italy

REFERENCES:
- [Derived] Carnevale L, Maffei A, Landolfi A, Grillea G, Carnevale D, Lembo G. Brain Functional Magnetic Resonance Imaging Highlights Altered Connections and Functional Networks in Patients With Hypertension. Hypertension. 2020 Nov;76(5):1480-1490. doi: 10.1161/HYPERTENSIONAHA.120.15296. Epub 2020 Sep 21. PMID 32951470